CLINICAL TRIAL: NCT03021850
Title: Comparison Between Different Therapeutical Modalities Associated to Hamstring Flexibility Training: Randomized Clinical Trial
Brief Title: Different Therapeutical Modalities Associated to Hamstring Flexibility Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Health Science of Porto Alegre (Other)
Responsible Party: Principal Investigator, Luis Henrique Telles da Rosa, Doctor, Federal University of Health Science of Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CAAE 52107115.7.0000.5345
Record Dates: First submitted 2017-01-06; First posted 2017-01-16 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Range of Motion, Articular
Keywords: Pliability; Cryotherapy; Hot temperature; Hyperthermia, induced; Randomized Controlled Trial; Hamstring muscles; Muscle stretching exercises
MeSH Terms: conditions — Hyperthermia

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Stretching associated with shortwave heating (Active Comparator): Applying deep heat through the shortwave equipment for 20 minutes, in coplanar application to the posterior part of the thigh associated with flexibility training of the hamstrings in the last 10 minutes of the session, performed by passive static stretching of the hamstring muscles in 10 repetitions of 30 seconds, with a 10 second pause between each repetition.
  Interventions: Procedure: Flexibility training with or without different thermal modalities
- Stretching associated with cryotherapy (Active Comparator): Cryotherapy application for 20 minutes, applied to the posterior part of the thigh associated with flexibility training of the hamstring muscles in the last 10 minutes of the session, performed by passive static stretching of the hamstring muscles, in 10 repetitions of 30 seconds , with a 10 second pause between each repetition.
  Interventions: Procedure: Flexibility training with or without different thermal modalities
- Stretching isolated (Other): The flexibility training of the hamstring muscles will be by passive static stretching of the hamstring muscles in 10 repetitions of 30-second , with a 10-second pause between each repetition.
  Interventions: Procedure: Flexibility training with or without different thermal modalities

INTERVENTIONS:
Procedure: Flexibility training with or without different thermal modalities — Flexibility training of the hamstring muscles by passive static stretching of the hamstring muscles in 10 30-second repetitions, with a 10-second pause between each repetition associated with or without short-wave heating or cryotherapy

SUMMARY:
The purpose of this study is to compare the acute effect of the use of different thermal modalities associated to the training of passive flexibility of the hamstring muscles in the amplitude of motion of the knee extension.

DETAILED DESCRIPTION:
Context: In the literature there is a disagreement of results and protocols regarding the use of thermal modalities associated with the training of flexibility of the hamstring muscles. Most studies on the subject, used the heat and cryotherapy prior to stretching these. Therefore, the investigators aimed to conduct an experimental study using the therapeutics term concomitant arrangements to passive static stretching these muscles.

Methods: Clinical trial randomized crossover, which will a sample of 42 subjects (healthy young men, aged 20 to 30 years). Were divided into 3 groups (Group 1 passive static stretching hamstrings, Group 2 heat + passive static stretching hamstrings and Group 3 cryotherapy + static stretching hamstrings passive) with 14 subjects each. Where the participants will control themselves, since all carry out the three interventions, only at different times. Each action will be performed every 7 days. Individuals will be subjected to active test of the range of motion of knee extension (goniometer) and hamstring muscle strength (dynamometer).

ELIGIBILITY:
Inclusion Criteria:

* Healthy men with knee extension range less than or equal to 160 degrees.

Exclusion Criteria:

* Have exercised in the last 48 hours before the intervention session;
* Previous neurological, muscular or articular disease that influences the performance of the training;
* Anterior lower limb surgery;
* Presence of painful symptoms or edema in the lower limbs;
* Hypersensitivity to ice or heat;
* Raynaud's syndrome;
* Loss of local thermal sensitivity;
* Have metallic implants;
* Use of cardiac pacemaker;
* Presence of malignant tumor;
* Arterial diseases;
* Deep venous thrombosis or phlebitis;
* Fever and inflammatory processes;
* Bleeding processes;
* Osteomyelitis;
* Epilepsy;
* Pulmonary and bone tuberculosis;
* Kidney or urinary tract infection;
* Cryoglobulinemia;

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2016-04-02 (Actual); Primary Completion 2017-02-10 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Change of Active Knee Extension Test | 3 weeks
  Active Knee Extension Test is performed in a standardised procedure and is measured in degrees.

SECONDARY OUTCOMES:
Change of Peak Torque of flexors and knee extensors | 3 weeks
  Peak torque of flexors and knee extensors is performed in an isokinetic dynamometer (Biodex system III), in a standardised procedure.
Change of Passive Resistance flexors and knee extensors | 3 weeks
  Passive Resistance of flexors and knee extensors is performed in an isokinetic dynamometer (Biodex system III), in a standardised procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Federal University of Health Science of Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Marek SM, Cramer JT, Fincher AL, Massey LL, Dangelmaier SM, Purkayastha S, Fitz KA, Culbertson JY. Acute Effects of Static and Proprioceptive Neuromuscular Facilitation Stretching on Muscle Strength and Power Output. J Athl Train. 2005 Jun;40(2):94-103. PMID 15970955
- [Result] Page P. Current concepts in muscle stretching for exercise and rehabilitation. Int J Sports Phys Ther. 2012 Feb;7(1):109-19. PMID 22319684
- [Result] Bandy WD, Irion JM, Briggler M. The effect of time and frequency of static stretching on flexibility of the hamstring muscles. Phys Ther. 1997 Oct;77(10):1090-6. doi: 10.1093/ptj/77.10.1090. PMID 9327823
- [Result] Bleakley CM, Costello JT. Do thermal agents affect range of movement and mechanical properties in soft tissues? A systematic review. Arch Phys Med Rehabil. 2013 Jan;94(1):149-63. doi: 10.1016/j.apmr.2012.07.023. Epub 2012 Aug 7. PMID 22885279
- [Result] Burke DG, Holt LE, Rasmussen R, MacKinnon NC, Vossen JF, Pelham TW. Effects of Hot or Cold Water Immersion and Modified Proprioceptive Neuromuscular Facilitation Flexibility Exercise on Hamstring Length. J Athl Train. 2001 Mar;36(1):16-19. PMID 12937509
- [Result] Brodowicz GR, Welsh R, Wallis J. Comparison of stretching with ice, stretching with heat, or stretching alone on hamstring flexibility. J Athl Train. 1996 Oct;31(4):324-7. PMID 16558418
- [Result] Draper DO, Castro JL, Feland B, Schulthies S, Eggett D. Shortwave diathermy and prolonged stretching increase hamstring flexibility more than prolonged stretching alone. J Orthop Sports Phys Ther. 2004 Jan;34(1):13-20. doi: 10.2519/jospt.2004.34.1.13. PMID 14964587
- [Result] Herbert RD, de Noronha M, Kamper SJ. Stretching to prevent or reduce muscle soreness after exercise. Cochrane Database Syst Rev. 2011 Jul 6;(7):CD004577. doi: 10.1002/14651858.CD004577.pub3. PMID 21735398
- [Result] Konrad A, Tilp M. Increased range of motion after static stretching is not due to changes in muscle and tendon structures. Clin Biomech (Bristol). 2014 Jun;29(6):636-42. doi: 10.1016/j.clinbiomech.2014.04.013. Epub 2014 May 10. PMID 24856792
- [Result] Rosario JL, Foletto A. Comparative study of stretching modalities in healthy women: heating and application time. J Bodyw Mov Ther. 2015 Jan;19(1):3-7. doi: 10.1016/j.jbmt.2013.12.003. Epub 2013 Dec 11. PMID 25603738
- [Result] Lim KI, Nam HC, Jung KS. Effects on hamstring muscle extensibility, muscle activity, and balance of different stretching techniques. J Phys Ther Sci. 2014 Feb;26(2):209-13. doi: 10.1589/jpts.26.209. Epub 2014 Feb 28. PMID 24648633
- [Result] Goncalves R, Gurjao AL, Jambassi Filho JC, Farinatti Pde T, Gobbi LT, Gobbi S. The acute effects of static stretching on peak force, peak rate of force development and muscle activity during single- and multiple-joint actions in older women. J Sports Sci. 2013;31(7):690-8. doi: 10.1080/02640414.2012.746727. Epub 2012 Dec 12. PMID 23234265
- [Result] Umegaki H, Ikezoe T, Nakamura M, Nishishita S, Kobayashi T, Fujita K, Tanaka H, Ichihashi N. Acute effects of static stretching on the hamstrings using shear elastic modulus determined by ultrasound shear wave elastography: Differences in flexibility between hamstring muscle components. Man Ther. 2015 Aug;20(4):610-3. doi: 10.1016/j.math.2015.02.006. Epub 2015 Mar 2. PMID 25795108
- [Result] Chen CH, Nosaka K, Chen HL, Lin MJ, Tseng KW, Chen TC. Effects of flexibility training on eccentric exercise-induced muscle damage. Med Sci Sports Exerc. 2011 Mar;43(3):491-500. doi: 10.1249/MSS.0b013e3181f315ad. PMID 20689450
- [Result] Nakano J, Yamabayashi C, Scott A, Reid WD. The effect of heat applied with stretch to increase range of motion: a systematic review. Phys Ther Sport. 2012 Aug;13(3):180-8. doi: 10.1016/j.ptsp.2011.11.003. Epub 2011 Dec 29. PMID 22814453
- [Result] Atamaz FC, Durmaz B, Baydar M, Demircioglu OY, Iyiyapici A, Kuran B, Oncel S, Sendur OF. Comparison of the efficacy of transcutaneous electrical nerve stimulation, interferential currents, and shortwave diathermy in knee osteoarthritis: a double-blind, randomized, controlled, multicenter study. Arch Phys Med Rehabil. 2012 May;93(5):748-56. doi: 10.1016/j.apmr.2011.11.037. Epub 2012 Mar 28. PMID 22459699
- [Result] Cornelius WL, Hands MR. The Effects of a Warm-up on Acute Hip Joint Flexibility Using a Modified PNF Stretching Technique. J Athl Train. 1992;27(2):112-4. PMID 16558145
- [Result] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Result] Opar DA, Williams MD, Timmins RG, Dear NM, Shield AJ. Knee flexor strength and bicep femoris electromyographical activity is lower in previously strained hamstrings. J Electromyogr Kinesiol. 2013 Jun;23(3):696-703. doi: 10.1016/j.jelekin.2012.11.004. Epub 2013 Jan 4. PMID 23290179
- [Result] Garrett CL, Draper DO, Knight KL. Heat distribution in the lower leg from pulsed short-wave diathermy and ultrasound treatments. J Athl Train. 2000 Jan;35(1):50-5. PMID 16558608